CLINICAL TRIAL: NCT02109224
Title: Phase I and Pharmacokinetic Study of Ibrutinib in HIV-Infected Patients With Relapsed or Refractory B-Cell Non-Hodgkin Lymphoma or Multiple Myeloma
Brief Title: Ibrutinib in Treating Relapsed or Refractory B-Cell Non-Hodgkin Lymphoma in Patients With HIV Infection
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Inadequate accrual rate
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2014-00707; NCI-2014-00707 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AMC-091 (Other: AIDS Malignancy Consortium); AMC-091 (Other: CTEP); U01CA121947 (NIH)
Record Dates: First submitted 2014-04-07; First posted 2014-04-09 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2015-04

CONDITIONS: Adult B Acute Lymphoblastic Leukemia; Chronic Lymphocytic Leukemia; Cutaneous B-Cell Non-Hodgkin Lymphoma; Extranodal Marginal Zone Lymphoma of Mucosa-Associated Lymphoid Tissue; HIV Infection; Intraocular Lymphoma; Multicentric Angiofollicular Lymphoid Hyperplasia; Nodal Marginal Zone Lymphoma; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Grade III Lymphomatoid Granulomatosis; Recurrent Adult Immunoblastic Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Small Lymphocytic Lymphoma; Refractory Chronic Lymphocytic Leukemia; Refractory Hairy Cell Leukemia; Refractory Plasma Cell Myeloma; Small Intestinal Lymphoma; Splenic Marginal Zone Lymphoma; Testicular Lymphoma; Waldenstrom Macroglobulinemia
MeSH Terms: conditions — Burkitt Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, B-Cell, Marginal Zone; HIV Infections; Intraocular Lymphoma; Multi-centric Castleman's Disease; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Leukemia, Hairy Cell; Multiple Myeloma; Waldenstrom Macroglobulinemia | interventions — ibrutinib

ARMS (1):
- Treatment (ibrutinib) (Experimental): Patients receive ibrutinib PO QD on days 1-28. Courses repeat every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Ibrutinib; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study

INTERVENTIONS:
Drug: Ibrutinib — Given PO
  Other Names: BTK Inhibitor PCI-32765; CRA-032765; PCI-32765
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase I trial studies the side effects and best dose of ibrutinib in treating B-cell non-Hodgkin lymphoma that has returned or does not respond to treatment in patients with human immunodeficiency virus (HIV) infection. Ibrutinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. It is not yet known whether it is safe for patients with HIV infection to receive ibrutinib while also taking anti-HIV drugs.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety and tolerability of single-agent ibrutinib in combination with antiretroviral therapy (ART) specifically with respect to ibrutinib metabolism in HIV-infected patients with relapsed or refractory B-cell neoplasms.

II. To determine the maximum tolerated dose (MTD) of ibrutinib in this setting.

SECONDARY OBJECTIVES:

I. To characterize ibrutinib pharmacokinetics in relation to ART-cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) interactions.

II. To describe toxicity in relation to plasma concentrations of ibrutinib and its main metabolite.

III. To estimate objective response rate, clinical benefit, times to tumor response and progression, and 6-month and 1-year progression-free and overall survival.

IV. To describe changes in HIV viral load, immunologic parameters, and Epstein-Barr virus (EBV) and human herpesvirus 8 (HHV-8) deoxyribonucleic acid (DNA) copy numbers in plasma and in peripheral blood mononuclear cells (PBMC) in relation to ibrutinib therapy.

OUTLINE: This is a dose-escalation study.

Patients receive ibrutinib orally (PO) once daily (QD) on days 1-28. Courses repeat every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Known HIV infection and histologically confirmed B-cell non-Hodgkin lymphoma or B-cell lymphoproliferative disease as follows, as defined by the World Health Organization classification:

  * Active B-cell non-Hodgkin lymphoma (cluster of differentiation [CD]20 positive or negative), chronic lymphocytic leukemia (CLL) or small lymphocytic lymphoma (SLL), or multiple myeloma that has relapsed, progressed, or been refractory to at least one regimen
  * Note: Patients with CLL, SLL, or mantle cell lymphoma (MCL) may only be enrolled in Stratum C
* At least 14 days between ibrutinib initiation and last cancer therapy; any number of prior cancer therapies is permitted; patients otherwise fit for blood or marrow transplantation (BMT) should receive second-line chemotherapy before considering enrollment
* Serologic documentation of HIV infection at any time prior to study entry, as evidenced by positive enzyme-linked immunosorbent assay (ELISA), positive Western blot, or any other federally approved licensed HIV test; alternatively, this documentation may include a record that another physician has documented that the participant has HIV infection based on prior ELISA and Western blot, or other approved diagnostic tests
* Participants must be on a stable antiretroviral regimen per current International Acquired Immunodeficiency Syndrome (AIDS) Society guidelines as follows, with no intention of changing the regimen within 8 weeks after ibrutinib initiation:

  * Choice of regimen: The specific antiretroviral agents are at physician discretion, and the use of investigational agents currently available on an expanded-access basis is allowed; use of experimental antiretroviral agents or those containing zidovudine (including Combivir and Trizivir) is prohibited
  * Patients with mantle cell lymphoma, CLL, or SLL must be on non-cytochrome P450, family 3, subfamily A, polypeptide 4 (CYPA3A4) modulating antiretroviral agents (Stratum C) to be eligible for this study
  * Patients may be switched to non-conflicting regimens in order to participate
  * Stability of regimen: With the exception of patients on zidovudine-based ART, any changes in antiretroviral regimen must be made at least 4 weeks prior to ibrutinib initiation; patients taking zidovudine-based ART must change to a non-zidovudine-based regimen at least 2 weeks prior to ibrutinib initiation; changes to ART therapy during the study may be made if medically necessary (e.g. toxicity, treatment failure)
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1 or 2 (Karnofsky >= 60%)
* Life expectancy >= 2 months
* Absolute CD4+ lymphocyte count: >= 75 cells/uL
* Absolute neutrophil count >= 750 cells/uL
* Platelets >= 50,000 cells/uL, or >= 30,000/uL if bone marrow is involved by malignancy
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.0 x institutional upper limit of normal (ULN), or =< 5.0 x ULN if attributable to malignancy
* Total bilirubin =< 2.0 x ULN, unless elevated bilirubin is attributable to Gilbert's syndrome or to HIV medications (e.g., indinavir, tenofovir, atazanavir)
* Creatinine clearance (CrCl) >= 40 mL/min (modified Cockcroft-Gault)
* All subjects must be screened for hepatitis B and C infection; subjects must either have no history of hepatitis B or C, or must meet the following criteria in order to e eligible:

  * Hepatitis B: Subjects infected with hepatitis B must receive anti-hepatitis B therapy; per Infectious Diseases Society of America (IDSA) and American Association for the Study of Liver Diseases (AASLD) guidelines, subjects that show no immunity, defined by the lack of hepatitis B surface antibody, and show evidence of chronic infection (i.e. hepatitis B surface antigen positive [HBsAg+], hepatitis B core antibody positive [HB core AB +], hepatitis B surface antibody negative [HBsAB-]) must be on anti-hepatitis B therapy throughout the study in order to be eligible; the exact hepatitis B therapy is at the discretion of the infection disease specialist or investigator; all patients diagnosed with hepatitis B must also meet the liver function test criteria listed above and have no evidence of cirrhosis; however, all patients who present with acute hepatitis B, or who show normal transaminases but are HBsAg+ and immunoglobulin M positive (IgM+) for hepatitis B core antigen, are ineligible
  * Hepatitis C: Subjects, who are hepatitis C antibody positive, with or without a positive hepatitis C ribonucleic acid (RNA) level, must meet the liver function test criteria listed above and have no evidence of cirrhosis; patients diagnosed with hepatitis C less than 6 months before enrollment will be considered to have acute hepatitis C and will be ineligible unless the hepatitis C viral load is undetectable
* Must in the opinion of the investigator be capable of complying with this protocol
* Patients may not begin protocol therapy within 7 days of major surgery or within 3 days of minor surgery
* Willingness of sexually active subjects to use adequate contraception; both men and women of child-bearing potential treated or enrolled on this study must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) before study entry, for the duration of study participation, and 4 months after completion of ibrutinib; men who only have sex with other men do not need to use contraception specifically for this study; (should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately)
* Ability to understand and willingness to sign a written informed consent document

Exclusion Criteria:

* Prior exposure to ibrutinib
* Receipt of any investigational agents within 14 days before the first dose of ibrutinib
* Failure to recover to baseline or Common Terminology Criteria for Adverse Events (CTCAE) =< grade 2 from clinically significant toxicities due to prior cancer therapies or to any investigational agents
* Active central nervous system involvement by malignancy; central nervous system disease that has been treated into remission is permitted; a chart note of the clinician's impression of lack of central nervous system (CNS) involvement is acceptable
* Patients who require concomitant treatment with CYP3A4/5 strong inhibitors or inducers OTHER than antiretroviral therapies for HIV

  * As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter product
  * A prednisone equivalent of < 20 mg daily is permitted in patients requiring chronic use; larger doses must be discontinued >= 7 days prior to ibrutinib initiation and are prohibited during study treatment
* Anticoagulation with warfarin or equivalent vitamin K antagonists within 28 days prior to starting ibrutinib and throughout the study
* Significant or uncontrolled intercurrent condition including, but not limited to:

  * Infection other than HIV, hepatitis B, or hepatitis C that is symptomatic or requires systemic treatment
  * Opportunistic infection within 60 days prior to enrollment
  * Currently active clinically significant cardiovascular disease such as uncontrolled arrhythmia, congestive heart failure, any class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification, or history of myocardial infection within 6 months prior to enrollment
  * History of stroke or intracranial hemorrhage within 6 months prior to enrollment
  * History of class B or class C cirrhosis, per the modified Child-Pugh classification
  * Psychiatric illness that would limit compliance
* Inability to swallow capsules whole, or disease significantly affecting gastrointestinal function and/or inhibiting small intestine absorption, such as malabsorption syndrome, small bowel resection, or poorly controlled inflammatory bowel disease affecting the small intestine
* History of prior malignancy, with the exception of the following:

  * Malignancy treated with curative intent and with no evidence of active disease present for more than 3 years prior to screening and felt to be at low risk for recurrence by treating physician
  * Adequately treated non-melanomatous skin cancer or lentigo maligna melanoma without current evidence of disease
  * Adequately treated cervical carcinoma in situ without current evidence of disease
  * Skin-limited Kaposi sarcoma that has not required systemic treatment within 6 months prior to study enrollment
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ibrutinib
* Pregnancy or breastfeeding; a pregnancy test must be performed within 7 days prior to ibrutinib initiation in women of childbearing potential; pregnant women are excluded; breastfeeding must be discontinued

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2014-09; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Incidence of toxicities assessed using National Cancer Institute (NCI) CTCAE version 4.0 | Up to 30 days
MTD of ibrutinib defined as the dose level in which no more than 1 out of 6 patients experiences a dose limiting toxicity assessed using NCI CTCAE version 4.0 | 28 days

SECONDARY OUTCOMES:
1-year OS | From start of study treatment to death, assessed at 6 months
  Probabilities of 1-year OS will be estimated with the Kaplan-Meier method and reported with 95% CI.
1-year PFS | From start of study treatment to relapse, progression, or death from any cause, whichever occurs first, assessed at 6 months
  Probabilities of 1-year PFS will be estimated with the Kaplan-Meier method and reported with 95% CI.
6-month overall survival (OS) | From start of study treatment to death, assessed at 6 months
  Probabilities of 6-month OS will be estimated with the Kaplan-Meier method and reported with 95% CI.
6-month progression free survival (PFS) | From start of study treatment to relapse, progression, or death from any cause, whichever occurs first, assessed at 6 months
  Probabilities of 6-month PFS will be estimated with the Kaplan-Meier method and reported with 95% CI.
Changes in EBV DNA copy numbers in plasma and in PBMCs in relation to ibrutinib therapy | Baseline to up to 30 days
  Changes will be analyzed with descriptive statistics. Where there are sufficient data, repeated measures analysis of variance will be used to assess the effect of ibrutinib on these parameters across time. If the data do not meet the assumptions of normality, the data will either be transformed or Friedman's test (i.e. non-parametric analogue to a repeated measures analysis of variance) will be used.
Changes in HHV-8 DNA copy numbers in plasma and in PBMCs in relation to ibrutinib therapy | Baseline to up to 30 days
  Changes will be analyzed with descriptive statistics. Where there are sufficient data, repeated measures analysis of variance will be used to assess the effect of ibrutinib on these parameters across time. If the data do not meet the assumptions of normality, the data will either be transformed or Friedman's test (i.e. non-parametric analogue to a repeated measures analysis of variance) will be used.
Changes in HIV viral load | Baseline to up to 30 days
  Changes will be analyzed with descriptive statistics. Where there are sufficient data, repeated measures analysis of variance will be used to assess the effect of ibrutinib on these parameters across time. If the data do not meet the assumptions of normality, the data will either be transformed or Friedman's test (i.e. non-parametric analogue to a repeated measures analysis of variance) will be used.
Changes in immunologic parameters | Baseline to up to 30 days
  Changes will be analyzed with descriptive statistics. Where there are sufficient data, repeated measures analysis of variance will be used to assess the effect of ibrutinib on these parameters across time. If the data do not meet the assumptions of normality, the data will either be transformed or Friedman's test (i.e. non-parametric analogue to a repeated measures analysis of variance) will be used.
Clinical benefit | Up to 30 days
  The proportion of patients achieving clinical benefit and their corresponding 95% CIs will be reported.
Objective response rate | Up to 30 days
  The proportion of patients achieving objective responses and their corresponding 95% confidence intervals (CIs) will be reported.
Pharmacokinetic (PK) parameters of ibrutinib in relation to ART-CYP3A4 interactions, including half-life (T1/2), oral clearance (CL/F), and area under the curve (AUC) | Course 1, day 8: pre-dose, 0.5, 1, 2, 4, 6, 8, and 24 hours
  Relevant individual PK parameters will be estimated using non-compartmental or compartmental PK methods. For each stratum, the PK variables will be tabulated and descriptive statistics (e.g., geometric means and coefficients of variation) calculated for each dose level. Pharmacokinetic parameters (i.e., T1/2, CL/F, and AUC) will be compared across relevant antiretroviral therapies using non-parametric statistical testing techniques.
Plasma concentrations of ibrutinib and its main metabolite | Up to 30 days
  Correlations with toxicity will be explored using non-parametric statistical testing techniques.
Time to tumor progression | Up to 30 days
  Time to tumor progression will be reported descriptively with medians and ranges.
Time to tumor response | From the first study treatment until documentation of first objective response, assessed up to 30 days
  Time to tumor response will be reported descriptively with medians and ranges.

CONTACTS AND LOCATIONS:
Overall Officials: Yvette Kasamon, Principal Investigator — AIDS Malignancy Consortium
Locations (7):
- United States (7):
  - UCLA Center for Clinical AIDS Research and Education, Los Angeles, California
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Siteman Cancer Center at Washington University, St Louis, Missouri
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Albert Einstein College of Medicine, The Bronx, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York